CLINICAL TRIAL: NCT01436513
Title: Phase 1, Open-Label, Randomized, Single-Dose, Crossover Bioequivalence And Food Effect Study For A New Formulation Of Premarin Compared With A Reference Tablet In Japanese Healthy Postmenopausal Women
Brief Title: A Study To Compare The Amount Of Premarin Components That Is Absorbed Into The Blood Of Japanese Healthy Postmenopausal Women Following Oral Administration Of Two Different Tablets Of Premarin Under Fast and Fed Conditions.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B2811002; 3117X3-1112
Record Dates: First submitted 2011-09-16; First posted 2011-09-19 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Primary Ovarian Insufficiency; Vaginitis; Metrorrhagia; Menopause
Keywords: bioequivalence; menometrorrhagia; climacteric disturbance; Estrogen Replacement Therapy; Estrogens Conjugated
MeSH Terms: conditions — Primary Ovarian Insufficiency; Vaginitis; Metrorrhagia

ARMS (4):
- A (Experimental): Premarin reference tablet as a single oral dose under fasted conditions
  Interventions: Drug: Premarin reference tablet (fasted)
- B (Experimental): Premarin new tablet as a single oral dose under fasted conditions
  Interventions: Drug: Premarin new tablet (fasted)
- C (Experimental): Premarin reference tablet as a single oral dose under fed conditions
  Interventions: Drug: Premarin reference tablet (fed)
- D (Experimental): Premarin new tablet as a single oral dose under fed conditions
  Interventions: Drug: Premarin new tablet (fed)

INTERVENTIONS:
Drug: Premarin reference tablet (fasted) — Premarin reference tablet, single dose, fasted conditions
  Arms: A
Drug: Premarin new tablet (fasted) — Premarin new tablet, single dose, fasted conditions
  Arms: B
Drug: Premarin reference tablet (fed) — Premarin reference tablet, single dose, fed conditions
  Arms: C
Drug: Premarin new tablet (fed) — Premarin new tablet, single dose, fed conditions
  Arms: D

SUMMARY:
The purpose of this study is to assess the bioequivalence and food effect for a new Premarin formulation compared with a Premarin reference tablet in Japanese healthy postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy postmenopausal women

Exclusion Criteria:

* History or current evidence of thrombophlebitis, thromboembolic disorders, or any coagulopathies.
* History or presence of malignancy or estrogen-dependent neoplasia. Subjects with a documented history of any malignancy, except for basal or squamous cell carcinoma of skin, which has been treated and fully resolved for a minimal 5 years.
* History or presence of benign or malignant liver tumor that developed during the use of oral contraceptives or other estrogen-containing products.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Plasma unconjugated estrone (baseline adjusted) pharmacokinetic parameter:Cmax | Day 1 to Day 4
Plasma unconjugated estrone (baseline adjusted) pharmacokinetic parameter:AUCall | Day 1 to Day 4
Plasma unconjugated equilin pharmacokinetic parameter:Cmax | Day 1 to Day 4
Plasma unconjugated equilin pharmacokinetic parameter:AUCall | Day 1 to Day 4

SECONDARY OUTCOMES:
Plasma unconjugated estrone (baseline adjusted) pharmacokinetic parameter:Tmax | Day 1 to Day 4
Plasma unconjugated estrone (baseline adjusted) pharmacokinetic parameter:AUClast | Day 1 to Day 4
Plasma unconjugated estrone (baseline adjusted) pharmacokinetic parameter:AUCinf | Day 1 to Day 4
Plasma unconjugated estrone (baseline adjusted) pharmacokinetic parameter:MRT | Day 1 to Day 4
Plasma unconjugated estrone (baseline adjusted) pharmacokinetic parameter:half-life | Day 1 to Day 4
Plasma unconjugated equilin pharmacokinetic parameter:Tmax | Day 1 to Day 4
Plasma unconjugated equilin pharmacokinetic parameter:AUClast | Day 1 to Day 4
Plasma unconjugated equilin pharmacokinetic parameter:AUCinf | Day 1 to Day 4
Plasma unconjugated equilin pharmacokinetic parameter:MRT | Day 1 to Day 4
Plasma unconjugated equilin pharmacokinetic parameter:half-life | Day 1 to Day 4
Plasma unconjugated estrone (baseline unadjusted) pharmacokinetic parameter:half-life | Day 1 to Day 4
Plasma unconjugated estrone (baseline unadjusted) pharmacokinetic parameter:Cmax | Day 1 to Day 4
Plasma unconjugated estrone (baseline unadjusted) pharmacokinetic parameter:Tmax | Day 1 to Day 4
Plasma unconjugated estrone (baseline unadjusted) pharmacokinetic parameter:AUClast | Day 1 to Day 4
Plasma unconjugated estrone (baseline unadjusted) pharmacokinetic parameter:AUCall | Day 1 to Day 4
Plasma unconjugated estrone (baseline unadjusted) pharmacokinetic parameter:MRT | Day 1 to Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Shinjyuku-ku, Tokyo, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2811002&StudyName=A%20Study%20To%20Compare%20The%20Amount%20Of%20Premarin%20Components%20That%20Is%20Absorbed%20Into%20The%20Blood%20Of%20Japanese%20Healthy%20Postmenopausal%20Women%20Followin